CLINICAL TRIAL: NCT06779058
Title: Retrospective and Prospective Multi-center Clinical Study of Magnetic Resonance Elastography in Evaluating Hepatic Fibrosis in Chronic Viral Hepatitis B
Brief Title: MR Elastography for Assessing Liver Fibrosis in Chronic Hepatitis B
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Deputy director of department of radology, Shengjing Hospital
Other Study IDs: ShengjingH CHB 2501
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Chronic Hepatitis B; Liver Fibrosis
Keywords: Magnetic resonance elastography; Liver stiffness; Antiviral therapy
MeSH Terms: conditions — Hepatitis B, Chronic; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective cohort of patients confirmed diagnosed with chronic hepatitis B: Patients aged ≥ 18 who have been diagnosed with chronic hepatitis B from Jan 2010 to Oct 2024
  Interventions: Device: MRE; Device: Liver biopsy
- Prospective follow-up cohort of patients confirmed diagnosed with chronic hepatitis B: Patients aged ≥ 18 who have been diagnosed with chronic hepatitis B, both treated and untreated from Aug 2022
  Interventions: Device: MRE; Device: Liver biopsy

INTERVENTIONS:
Device: MRE — All imaging studies were performed by using a 1.5T/3.0-T MRI system
Device: Liver biopsy — Liver biopsy are performed by well-trained pathologists in accordance with standard operating procedures.

SUMMARY:
How to construct a non-invasive, accurate, and convenient method to evaluate the severity of liver fibrosis (LF) is an important general problem in the management of patients with chronic hepatitis B (CHB). We plan to investigate the ability of magnetic resonance elastography (MRE) to grade fibrosis in chronic hepatitis B and apply to clinical longitudinal follow-up.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is the most prevalent chronic viral infection worldwide, affecting 254 million people and resulting in 1.2 million new infections annually . Chronic hepatitis B (CHB) is strongly associated with liver fibrosis, cirrhosis, hepatocellular carcinoma, and death. Patients with chronic hepatitis C (CHC) can achieve an overall cure rate of more than 95% after 12 weeks of treatment with direct-acting antiviral agent (DAA). However, patients with chronic hepatitis B still need long-term management due to the complexity and persistence of their disease. Therefore, rapid, stable and accurate assessment of the disease status of hepatitis B patients and clear classification of liver fibrosis are of great significance for clinical management of chronic hepatitis B patients.

Meanwhile, Antiviral therapy can significantly slow liver disease progression and improve long-term survival in CHB patients. Treatment is only recommended for CHB adults when histological evidences ≥ F2; evidence of F4 based on clinical criteria; HBV DNA > 2000 IU/mL with ALT > ULN (Men: 30 U/L, Women: 19 U/L); or persistent ALT abnormality. For treated patients, imaging and clinical indicators are monitored every six months during the first year, then annually. For untreated patients, monitoring is conducted on an annual basis . However, these current tests often fail to reflect pathological changes in real-time, as they tend to lag behind actual disease progression. Therefore, finding an effective method for regular follow-up is also essential for both treated and untreated patients.

The current diagnostic gold standard, liver biopsy, has limitations due to its invasive nature, sampling error, complications, and high cost, making it impractical for evaluating liver fibrosis and longitudinal monitoring in CHB patients. There is an urgent need for noninvasive evaluation of liver fibrosis and antiviral treatment efficacy. Magnetic resonance elastography (MRE) has shown promise in assessing liver fibrosis and necroinflammation in CHB patients. At present, there are few studies on CHB, all of which are single-center studies. The reported cut-off point is not uniform, which is generally lower than the international standard, and whether 2D/3D MRE affects the threshold are inconsistent. Therefore, a multi-center clinical study on the evaluation of CHB fibrosis based on MRE and its application in clinical longitudinal follow-up need to be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Confirmed CHB (laboratory, imaging and clinical tests)
* MRE within 6 months before and after liver biopsy
* Treatment-naïve
* Child-Pugh Grade A (<7 points)
* Written informed consent in prospective follow-up cohort

Exclusion Criteria:

* Patients with liver malignant tumor
* Chronic hepatitis due to other causes (such as alcoholic hepatitis)
* CHB combined with hepatitis C, hepatitis D, or HIV
* Patients with biliary tract diseases
* Contraindications of MRE examination, MRE failure
* Poor pathological effect

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Organize paticipating units to collect standard-of-care data including radiological and clinical data. Patients diagnosed with CHB who received liver biopsy and MRE should be enrolled.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the features of MRE for grading fibrosis in chronic hepatitis B. | 6 months
  WIth liver biopsy as reference standand, the diagnostic perforemace (accuracy) for fibrosis of MRE was assessed.

SECONDARY OUTCOMES:
The efficacy of grading liver fibrosis in CHB patients evaluated by MRE superior to TE and serological indicators (APRI, FIB-4). | 6 months
  WIth liver biopsy as reference standand, the efficacy of MRE, TE and serological indicators (APRI, FIB-4) in evaluating the classification of liver fibrosis were compared.
The excellent ability of MRE as a non-invasive biomarker for longitudinal monitoring in CHB patients. | 12 months
  WIth QIBA Profile: Magnetic Resonance Elastography of the Liver as reference standand, changes in MRE and liver histology or clinical indicators during follow-up were investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided